CLINICAL TRIAL: NCT03041948
Title: Evaluating Pain Outcomes of Caudal vs Ilioinguinal Nerve Block in Children Undergoing Hernia Repair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alberta Children's Hospital (Other)
Collaborators: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Bryce Weber, Pediatric Urologist, Alberta Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: REB15-0434
Record Dates: First submitted 2017-02-01; First posted 2017-02-03 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Hernia, Inguinal; Pain, Postoperative
Keywords: Inguinal hernia; Caudal nerve block; Ilioinguinal nerve block; Pain
MeSH Terms: conditions — Hernia, Inguinal; Pain, Postoperative; Pain | interventions — Acetaminophen; Sevoflurane; Remifentanil; Propofol; Morphine; Ondansetron; Dexamethasone; Ketorolac

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Caudal-epidural nerve block (Active Comparator): All patients will receive acetaminophen (15mg/kg) within one hour of induction of anesthesia. Inhalation induction of anesthesia will be performed with sevoflurane in 100% O2. A single dose of up to 2-4 mg/kg of propofol and Remifentanil 0.5-1mcg/kg will be given prior insertion of a laryngeal mask airway or endotracheal tube. Anesthesia will be maintained with Propofol and Remifentanil (2.5mcg/ml) which will be started at 300 mcg/kg/min and titrated to effect. If necessary additional boluses of Propofol (1mg/kg) and/or Remifentanil (0.5-1mcg/kg) and/or Morphine 0.05mg/kg boluses IV will be administered. Ondansetron (0.1mg/kg) and Dexamethasone (0.15mg/kg) will be given as antiemetic prophylaxis for all patients. Ketorolac 0.3mg/kg will be given to each patient. The CE group will receive an US-confirmed CE nerve block with 0.8 mL/kg of 0.2% ropivacaine (maximum 15 mL).
  Interventions: Procedure: Caudal-epidural nerve block; Drug: Acetaminophen; Drug: Sevoflurane; Drug: Remifentanil; Drug: Propofol; Drug: Morphine; Drug: Ondansetron; Drug: Dexamethasone; Drug: Ketorolac
- ilioinguinal/iliohypogastric nerve block (Experimental): All patients will receive acetaminophen (15mg/kg) within one hour of induction of anesthesia. Inhalation induction of anesthesia will be performed with sevoflurane in 100% O2. A single dose of up to 2-4 mg/kg of propofol and Remifentanil 0.5-1mcg/kg will be given prior insertion of a laryngeal mask airway or endotracheal tube. Anesthesia will be maintained with Propofol and Remifentanil (2.5mcg/ml) which will be started at 300 mcg/kg/min and titrated to effect. If necessary additional boluses of Propofol (1mg/kg) and/or Remifentanil (0.5-1mcg/kg) and/or Morphine 0.05mg/kg boluses IV will be administered. Ondansetron (0.1mg/kg) and Dexamethasone (0.15mg/kg) will be given as antiemetic prophylaxis for all patients. Ketorolac 0.3mg/kg will be given to each patient. The IIG/IHG group will receive a unilateral US guided IIG/IHG with 0.4mL/kg of ropivacaine 0.2% (max 12 mL).
  Interventions: Procedure: Ilioinguinal/iliohypogastric nerve block; Drug: Acetaminophen; Drug: Sevoflurane; Drug: Remifentanil; Drug: Propofol; Drug: Morphine; Drug: Ondansetron; Drug: Dexamethasone; Drug: Ketorolac

INTERVENTIONS:
Procedure: Ilioinguinal/iliohypogastric nerve block — See arm description
  Arms: ilioinguinal/iliohypogastric nerve block
Procedure: Caudal-epidural nerve block — See arm description
  Arms: Caudal-epidural nerve block
Drug: Acetaminophen — See arm description
Drug: Sevoflurane — See arm description
Drug: Remifentanil — See arm description
Drug: Propofol — See arm description
Drug: Morphine — See arm description
Drug: Ondansetron — See arm description
Drug: Dexamethasone — See arm description
Drug: Ketorolac — See arm description

SUMMARY:
Surgical intervention to treat a inguinal hernia is a very common pediatric surgical procedure, often performed using an inguinal incision. Children who undergo hernia repair can suffer from a significant degree of discomfort postoperatively. The investigators are evaluating the effectiveness of an ultrasound guided caudal-epidural (CE) block to an US guided ilioinguinal/iliohypogastric (IIG/IHG) nerve block in achieving post operative analgesia following a hernia repair. It is hypothesized that US guided IIG/IHG nerve block leads to more effective pain control post-operatively while in hospital relative to an US guided CE block for inguinal hernia surgery.

DETAILED DESCRIPTION:
Surgical intervention to treat a inguinal hernia is a very common pediatric surgical procedure, often performed using an inguinal incision. Children who undergo hernia repair can suffer from a significant degree of discomfort postoperatively. A multimodal pain management approach including medications such as acetaminophen, non-steroidal anti-inflammatory drugs and opioids have traditionally been used in combination with a regional anesthetic technique. Regional anesthetic techniques include surgical infiltration of local anesthetic, caudal-epidural (CE) block or an ilioinguinal/iliohypogastric (IIG/IHG) nerve block.

Regional anesthetic techniques such as CE and ultrasound (US) guided IIG/IHG are well-established methods shown to reduce the use of intraoperative anesthetics and the need post operative rescue analgesia. Traditionally, IIG/IHG nerve blocks were completed using a landmark-based approach but due to unpredictable block results with failure rates over 30% and potentially serious complications such as unintentional intraperitoneal injection, many anesthesiologists preferred the more reliable CE technique. However, while the CE provides excellent intraoperative anesthesia it provides short duration of post-operative analgesia (4-6 hours) and can be associated with lower limb motor block and urinary retention. Recent literature has demonstrated that an US guided IIG/IHG can be completed with smaller volume of local anesthetic with a success rate of up to 100% with low risk of complications. Furthermore there is evidence to suggest that it provides an increased duration of postoperative analgesia for pediatric patients undergoing groin surgery. Finally, two publications retrospectively reviewing complications in over 45000 regional anesthetic blocks suggest that US guided peripheral nerve blocks (e.g., IIG/IHG) should be favoured over neuraxial techniques such as epidural and caudal anesthetics due to the risk-benefit profile. A recent meta-analysis comparing IIG/IIH block to the CE block in children notes that additional comparative studies are required as previous studies comparing these two techniques have many methodological limitations including small sample sizes, using blind (non-US guided) regional anesthetic techniques and grouping patients undergoing various surgical procedures (e.g., orchiopexy and hernia repair) despite significant differences in recovery pain profiles.

The investigators are proposing to complete a prospective randomized single-blinded non-inferiority study to evaluate and compare the effectiveness of an US guided CE block to an US guided IIG/IHG nerve block in achieving post operative analgesia following a hernia repair. Currently, a number of Pediatric Anesthesiologists at the Alberta Children's Hospital do not routinely complete IIG/IIH or CE blocks under ultrasound guidance. As part of this study investigators hope to provide necessary knowledge (sonoanatomy, technique) and offer supervised clinical training to anesthesiologists who are interested in participating in the study. While a hernia repair remains a common procedure, no studies have compared the use of US guided CE to US guided IIG/IHG. The aim of this study is to establish non-inferiority in post-operative pain while in hospital as assessed through the Face, Leg, Activity, Cry, Consolability (FLACC) scale for the US guided IIG/IHG as compared to US guided CE following hernia repair surgery. Secondary objectives will assess for group differences in need for rescue analgesia in hospital, analgesia administered at home, and postoperative pain measures within 24 hours post hospital discharge.

Investigators hypothesize that a US guided IIG/IHG nerve block leads to non-inferior objectively measured FLACC pain scores (≤ 1 point on FLACC scale) post-operatively while in hospital relative to an US guided CE block for inguinal hernia surgery.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children (ASA I and II) between the ages of 6 months and 4 years presenting for elective hernia repair who are scheduled for day stay only.

Exclusion Criteria:

* Patients with a history of clinically important renal, hepatic, cardiac, or neurological conditions and those with a history of allergic reactions to local anesthetics, bleeding diatheses, coagulopathy, and spinal abnormality such as a sacral dimple will be excluded.

Ages: 6 Months to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 88 (Estimated)
Dates: Start 2015-09-01 (Actual); Primary Completion 2018-09-01 (Estimated); Study Completion 2018-09-01 (Estimated)

PRIMARY OUTCOMES:
Post-operative pain | Immediately following the procedure
  Evaluated through the use of the Face, Legs, Activity, Cry, Consolability (FLACC) pain score by a nurse or research assistant blinded to the anesthetic technique. The FLACC scale is out of 10 and is used in children who have difficulty verbalizing pain and in sleeping children (regardless of age).
Post-operative pain | 15 minutes post-operatively
  Evaluated through the use of the Face, Legs, Activity, Cry, Consolability (FLACC) pain score by a nurse or research assistant blinded to the anesthetic technique. The FLACC scale is out of 10 and is used in children who have difficulty verbalizing pain and in sleeping children (regardless of age).
Post-operative pain | 30 minutes post-operatively
  Evaluated through the use of the Face, Legs, Activity, Cry, Consolability (FLACC) pain score by a nurse or research assistant blinded to the anesthetic technique. The FLACC scale is out of 10 and is used in children who have difficulty verbalizing pain and in sleeping children (regardless of age).
Post-operative pain | 60 minutes post-operatively
  Evaluated through the use of the Face, Legs, Activity, Cry, Consolability (FLACC) pain score by a nurse or research assistant blinded to the anesthetic technique. The FLACC scale is out of 10 and is used in children who have difficulty verbalizing pain and in sleeping children (regardless of age).
Post-operative pain | 120 minutes post-operatively
  Evaluated through the use of the Face, Legs, Activity, Cry, Consolability (FLACC) pain score by a nurse or research assistant blinded to the anesthetic technique. The FLACC scale is out of 10 and is used in children who have difficulty verbalizing pain and in sleeping children (regardless of age).

SECONDARY OUTCOMES:
Post-operative pain | 24 hours post-operatively
  Patients will be contacted 24 hours following their surgery to complete the parents' postoperative pain measure (PPPM). The PPPM is a well-established post-operative pain assessment tool with high inter-rater reliability and construct validity that has been designed specifically for use by parents in the post-operative care of their children. The measure includes 15 items scored between 0 and 1. The questionnaire will be completed over the telephone within 24 hours of the patient's surgery.
Total ibuprofen consumption | Up to 24 hours post-operatively
  Evaluated and compiled through anesthesia notes, post-operative nursing care notes and parental telephone follow-up
Total acetaminophen consumption | Up to 24 hours post-operatively
  Evaluated and compiled through anesthesia notes, post-operative nursing care notes and parental telephone follow-up

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Alberta Children's Hospital, Calgary, Alberta
  - Royal University Hospital/University of Saskatchewan, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Verghese ST, Hannallah RS. Acute pain management in children. J Pain Res. 2010 Jul 15;3:105-23. doi: 10.2147/jpr.s4554. PMID 21197314
- [Background] Koo BN, Hong JY, Song HT, Kim JM, Kil HK. Ultrasonography reveals a high prevalence of lower spinal dysraphism in children with urogenital anomalies. Acta Anaesthesiol Scand. 2012 May;56(5):624-8. doi: 10.1111/j.1399-6576.2011.02612.x. Epub 2012 Feb 16. PMID 22338610
- [Background] Weintraud M, Marhofer P, Bosenberg A, Kapral S, Willschke H, Felfernig M, Kettner S. Ilioinguinal/iliohypogastric blocks in children: where do we administer the local anesthetic without direct visualization? Anesth Analg. 2008 Jan;106(1):89-93, table of contents. doi: 10.1213/01.ane.0000287679.48530.5f. PMID 18165559
- [Background] Jagannathan N, Sohn L, Sawardekar A, Ambrosy A, Hagerty J, Chin A, Barsness K, Suresh S. Unilateral groin surgery in children: will the addition of an ultrasound-guided ilioinguinal nerve block enhance the duration of analgesia of a single-shot caudal block? Paediatr Anaesth. 2009 Sep;19(9):892-8. doi: 10.1111/j.1460-9592.2009.03092.x. Epub 2009 Jul 13. PMID 19627532
- [Background] Abdellatif AA. Ultrasound-guided ilioinguinal/iliohypogastric nerve blocks versus caudal block for postoperative analgesia in children undergoing unilateral groin surgery. Saudi J Anaesth. 2012 Oct-Dec;6(4):367-72. doi: 10.4103/1658-354X.105868. PMID 23493806
- [Background] Ecoffey C, Lacroix F, Giaufre E, Orliaguet G, Courreges P; Association des Anesthesistes Reanimateurs Pediatriques d'Expression Francaise (ADARPEF). Epidemiology and morbidity of regional anesthesia in children: a follow-up one-year prospective survey of the French-Language Society of Paediatric Anaesthesiologists (ADARPEF). Paediatr Anaesth. 2010 Dec;20(12):1061-9. doi: 10.1111/j.1460-9592.2010.03448.x. PMID 21199114
- [Background] Polaner DM, Taenzer AH, Walker BJ, Bosenberg A, Krane EJ, Suresh S, Wolf C, Martin LD. Pediatric Regional Anesthesia Network (PRAN): a multi-institutional study of the use and incidence of complications of pediatric regional anesthesia. Anesth Analg. 2012 Dec;115(6):1353-64. doi: 10.1213/ANE.0b013e31825d9f4b. Epub 2012 Jun 13. PMID 22696610
- [Background] Shanthanna H, Singh B, Guyatt G. A systematic review and meta-analysis of caudal block as compared to noncaudal regional techniques for inguinal surgeries in children. Biomed Res Int. 2014;2014:890626. doi: 10.1155/2014/890626. Epub 2014 Aug 5. PMID 25162033
- [Background] von Baeyer CL, Spagrud LJ. Systematic review of observational (behavioral) measures of pain for children and adolescents aged 3 to 18 years. Pain. 2007 Jan;127(1-2):140-50. doi: 10.1016/j.pain.2006.08.014. Epub 2006 Sep 25. PMID 16996689
- [Background] Merkel SI, Voepel-Lewis T, Shayevitz JR, Malviya S. The FLACC: a behavioral scale for scoring postoperative pain in young children. Pediatr Nurs. 1997 May-Jun;23(3):293-7. PMID 9220806
- [Background] Chambers CT, Finley AG, McGrath PJ, Walsh TM. The parents' postoperative pain measure: replication and extension to 2-6-year-old children. Pain. 2003 Oct;105(3):437-443. doi: 10.1016/S0304-3959(03)00256-2. PMID 14527704
- [Background] Cole J, Shepherd M, Young P. Intranasal fentanyl in 1-3-year-olds: a prospective study of the effectiveness of intranasal fentanyl as acute analgesia. Emerg Med Australas. 2009 Oct;21(5):395-400. doi: 10.1111/j.1742-6723.2009.01216.x. PMID 19840089